CLINICAL TRIAL: NCT02005406
Title: Efficacy and Safety of the WEI Nasal Jet
Brief Title: Testing the Efficacy and Safety of the WEI Nasal Jet
Acronym: WNJ
Status: Completed | Type: Observational
Sponsor: Zeyong Yang (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor-Investigator, Zeyong Yang, Shanghai Jiaotong University, Fudan University
Organization: Fudan University (Other)
Other Study IDs: Wei JET
Record Dates: First submitted 2013-07-03; First posted 2013-12-09 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2013-12

CONDITIONS: Complication of Surgical Procedure
Keywords: Wei JET

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — •Patients receiving various types of surgeries under sedation, especially for procedures of colonoscopy, upper gastrointestinal endoscopy, endoscopic retrograde cholangiopancreatography (ERCP) cystoscopy and other brief surgeries you are interested in the study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- wei group and control group: wei group(n=25) and control group(n=24)
  Interventions: Device: Experimental group and control groupl

INTERVENTIONS:
Device: Experimental group and control groupl — JET
  Other Names: WEI; Control

SUMMARY:
Testing the efficacy and safety of the WEI Nasal Jet.

DETAILED DESCRIPTION:
This is only initial thought and suggestions from the inventor Dr. Huafeng Wei. Principal investigator from each medical center interested in testing this new device should design their own clinical trials based on patient population and their own ideas for clinical trials. Just remind you that patient safety is number one and try all efforts to minimize patient risks during your clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving various types of surgeries under sedation, especially for procedures of colonoscopy, upper gastrointestinal endoscopy, endoscopic retrograde cholangiopancreatography (ERCP) cystoscopy and other brief surgeries you are interested in the study.

Exclusion Criteria:

* Patients with coagulopathy and tendency of nose bleeding.
* Patients with any diagnosed cardiac diseases (e.g. cardiac failure, angina, MI, cardiac arrhythmia. etc.)
* Patients with any diagnosed pulmonary disease (e.g. asthma, COPD, pulmonary embolism, pulmonary edema etc.)
* Pregnant patients
* Patients with liver failure
* Patients with kidney failure

Ages: 22 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Suggested patient inclusion criteria:
  Patients receiving various types of surgeries under sedation, especially for procedures of colonoscopy, upper gastrointestinal endoscopy, endoscopic retrograde cholangiopancreatography (ERCP) cystoscopy and other brief surgeries you are interested in the study.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
lowest SaO2 in Wei JET group | 2 second
  Compare with Control group,there was no significant difference in lowest SaO2 in Wei JET group.

CONTACTS AND LOCATIONS:
Overall Officials: Zeyong Yang, MD, Ph.D, Principal Investigator — Shanghai Jiao Tong University School of Medicine

REFERENCES:
- [Derived] Yang ZY, Meng Q, Xu YH, Wang JW, Yu DS, Wei HF. Supraglottic jet oxygenation and ventilation during colonoscopy under monitored anesthesia care: a controlled randomized clinical trial. Eur Rev Med Pharmacol Sci. 2016;20(6):1168-73. PMID 27049273